CLINICAL TRIAL: NCT05589623
Title: Adding the Copenhagen Adductor Exercise to Standard Groin Injury Rehabilitation: A Randomized Controlled Trial
Brief Title: The Effectiveness of the Copenhagen Adduction Exercise on Soccer Players With Groin Pain or Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Ahmed Alsirhani, Principal Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2023-03-011
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Groin Injury
Keywords: Copenhagen Adduction Exercise; Eccentric Hip Adduction Strength; Groin injury, groin pain; Soccer. athletes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copenhagen adduction exercise (Experimental): The CAE is a body-weight exercise that mainly works the groin and hip adductors. It has a significant eccentric component, meaning the muscles work while lengthening. The CAE is a simple isolated eccentric exercise that does not require special equipment. Due to the heaviness and the high dynamic demands of CAE, a modified progressive Copenhagen adduction (MPCA) program has been created. The MPCA exercise was adapted from the original CAE to lessen the risk of delayed onset muscle soreness (DOMS) and facilitate high participant compliance. An experienced physical therapist will include the MPCA in the usual rehabilitation program for eight weeks, twice weekly. Sessions will last between 30 and 120 minutes.
  Interventions: Other: Copenhagen adduction exercise
- Usual rehabilitation program (Active Comparator): The rehabilitation program will be an active exercise based on the available literature and considers the clinical experience in managing groin injuries. An experienced physical therapist will supervise the rehabilitation program for two sessions weekly for eight weeks, with difficulty and volume progressing incrementally. Sessions will last between 30 and 120 minutes.
  Interventions: Other: Usual rehabilitation program

INTERVENTIONS:
Other: Copenhagen adduction exercise — The CAE is a progressive eccentric training program that enhances hip adduction. The fact that exercises are done with a partner and do not require special equipment makes them more useful in a team setting. The MPCA program, adapted from the original CAE, included six progressive levels for eight weeks, beginning with an assisted isometric adduction hold (level 1) and progressing incrementally to a complete CAE as the original exercise (level 6). The progression in levels will depend on a pain score ≤ 4/10 numeric rating scale (NRS) in the adductor squeeze test and post-session DOMS score ≤ 4/10 NRS.
  Arms: Copenhagen adduction exercise
Other: Usual rehabilitation program — The usual rehabilitation program will include leg swings extension/flexion, leg swings abduction/adduction, standing hip circles, isometric standing hip adduction using elastic bands, stretching exercises, balance training on a wobble board, and single leg coordination exercises. Difficulty and volume are progressing incrementally.
  Arms: Usual rehabilitation program

SUMMARY:
Groin injuries are among the three most common and time-consuming injuries in soccer, accounting for 19% of all injuries, with 0.1-2.1 injuries per 1000 hours of play. The Copenhagen Adduction Exercise (CAE) has been showing promising results in improving Eccentric Hip Adduction Strength (EHADS), leading to reducing the risk of groin pain and injury. This clinical trial aims to evaluate the effects of CAE on adductors strength, hip joint range of motion (ROM), and Patient-reported outcome measures among athletes with groin pain or injury.

The main question it aims to answer is:

Does the CAE improve EHAD strength, hip joint ROM, and patient-reported outcome measures among soccer players with groin pain or injury?

Researchers will assess the participants' pre and post-intervention to determine the effects of CAE on adductors strength, hip joint ROM, and Patient-reported outcome measures.

DETAILED DESCRIPTION:
Study design: A Double-Blinded Randomized Controlled Trial.

Researchers will allocate a specific number for each participant for randomization. Then, an online website will be applied to randomize these numbers into two groups, intervention and control groups. An independent person not involved in the study will allocate the participants using concealed opaque envelopes.

Study setting:

This study will be held at different physical therapy and rehabilitation clinic, ministry of health, Saudi Arabia

Recruitment and study population:

Participants will be recruited from physical therapy outpatient clinics in the South region.

Participants will be recruited and randomized into two groups, intervention (CAE) and control. Participants assigned to the intervention group will receive the CAE in addition to the regular physical therapy rehabilitation program for eight weeks. Due to the heaviness and the high dynamic demands of CAE, a modified progressive Copenhagen adduction (MPCA) program has been created. The MPCA was adapted from the original CAE to lessen the risk of delayed onset muscle soreness (DOMS) and facilitate high participant compliance.

Participants assigned to the control group will receive the same physical therapy rehabilitation program as the intervention group except for the CAE.

Time plan of the study:

Recruitment is expected to commence in January 2023 and conclude in April 2023. After completing the recruitment process, data will be collected for eight weeks. After the last inclusion, the intervention will continue for eight weeks.

Assessment:

An experienced physiotherapist, blinded to the study, will perform all assessments to guarantee that the tests are consistent and that the process is standardized. Assessments will be at baseline and post-intervention. The duration between the baseline assessment and the start of the intervention should not exceed two weeks. After the assessment, every participant will receive the proper group intervention according to his/her randomization. Participants will be told not to reveal their group assignments to the assessor during the study period.

Demographic variables and descriptive:

The investigators will document the following variables: age, sex, height, BMI, Sports level, duration of symptoms, and location of symptoms as recommended by the minimum reporting criteria for clinical research on groin pain in athletes.

Sample size estimation:

The sample size calculation for this study was performed using G*Power software (v. 3.1, Heinrich-Heine-Universität, Düsseldorf, Germany), with an alpha level of 0.05 and a power (1-β) of 80%. Based on a previous study examining the effects of exercise therapy on adductor-related groin pain in athletes, it required 15 participants per group to detect an expected between-group difference of 0.15 Nm/kg and a standard deviation (SD) of 0.54 Nm/kg.

Statistical analysis:

All analyses will be performed using the Statistical Package for the Social Sciences version 27. The study's findings will be presented following the Consolidated Standards of Reporting Trials (CONSORT). Shapiro-Wilk test will be used to test for normality. The statistical analysis test will be carried out based on the collected data. Demographic data will be presented as mean and standard deviation. The suggested statistical analysis measure will be the repeated measures analysis of variance (ANOVA), calculated for each dependent variable. Each repeated measure ANOVA will have one within factor (test: pre and post) and one between factor (group: training and control). Results will be significant at P value <0.05 and a Confidence Interval (CI) of 95%. A statistician will be consulted for further correction after data collection.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players aged between 18 to 40 years.
* They have groin pain or injury within two months during sports.
* Pain or tenderness on palpation of adductors in clinical examination.
* Pain on resisted hip adduction movement in clinical examination.
* Desire to continue the sport at the same level.

Exclusion Criteria:

* Groin pain or injury not involving the adductors on clinical examination.
* They have any clinical finding indications of femoral or inguinal hernia.
* Evidence of prostatitis, chronic urinary tract disease.
* Evidence of hip joint osteoarthritis or hip joint disease.
* Bursitis of the hip or groin region.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Change in eccentric hip adduction strength from baseline | At the end of the intervention sessions (8 weeks)
  A portable hand-held dynamometer (microFET2) will be used for the test. A blind physiotherapist will perform pre and post-testing. Each patient's affected leg will be tested. The examiner will position the hand-held dynamometer 5 cm proximal to the most prominent part of the medial malleolus. Eccentric hip adduction strength will be measured in a break test with the patient in a side-lying position, with the leg being tested in a straight position. The participant will perform a 3-5 second isometric maximum voluntary contraction against the dynamometer before the physiotherapist performs a contraction break to determine the eccentric hip adduction strength. The patient will complete one practice trial before three maximal tests are performed, with the best result recorded. The standardized command by the examiner will be "go ahead-push-push-push-push-push." Leg length will be used to calculate torque and be adjusted to body mass (Nm/kg).
Change in hip joint range of motion measures from baseline | At the end of the intervention sessions (8 weeks)
  Hip joint ROM can be reliably assessed using a goniometer. The assessor will perform an internal and external hip joint range of motion testing with the subject supine and the hip and knee in 90 degrees of flexion pre-and post-testing will be performed. An assistant will be used to ensure that the hip and knee remain in their proper positions. The affected leg will be rotated to the maximum range of passive internal rotation (IR), external rotation (ER), and abduction movement (ABD). The standard goniometer will be used to make the measurements, and the testing period will be approximately ten minutes.

SECONDARY OUTCOMES:
Change in the Copenhagen Hip and Groin Outcome Score | At the end of the intervention sessions (8 weeks)
  The Copenhagen Hip and Groin Outcome Score (HAGOS) was created as a patient-reported outcome questionnaire, primarily targeting young-aged to middle-aged, physically active individuals with long-standing hip and groin pain. HAGOS, was existed for specifically assessing those reporting groin pain. The HAGOS comprises six subscales that assess pain, symptoms, physical function in daily life, physical function in sport and recreation, participation in physical activities, and hip and/or groin-related quality of life (QOL). Scores for each subscale range from 0 (extreme hip/groin problems) to 100 (no hip/groin problems). The Arabic version of HAGOS has been recommended for assessing symptoms, activity limitations, participation restrictions, and quality of life in physically active, young, middle-aged patients with hip and/or groin pain.

CONTACTS AND LOCATIONS:
Overall Officials: Qassim Muaidi, Professor, Study Chair — Imam Abdulrahman Bin Faisal University
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delahunt E, Thorborg K, Khan KM, Robinson P, Holmich P, Weir A. Minimum reporting standards for clinical research on groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):775-81. doi: 10.1136/bjsports-2015-094839. PMID 26031644
- [Background] Haroy J, Thorborg K, Serner A, Bjorkheim A, Rolstad LE, Holmich P, Bahr R, Andersen TE. Including the Copenhagen Adduction Exercise in the FIFA 11+ Provides Missing Eccentric Hip Adduction Strength Effect in Male Soccer Players: A Randomized Controlled Trial. Am J Sports Med. 2017 Nov;45(13):3052-3059. doi: 10.1177/0363546517720194. Epub 2017 Aug 14. PMID 28806100
- [Background] Ishoi L, Sorensen CN, Kaae NM, Jorgensen LB, Holmich P, Serner A. Large eccentric strength increase using the Copenhagen Adduction exercise in football: A randomized controlled trial. Scand J Med Sci Sports. 2016 Nov;26(11):1334-1342. doi: 10.1111/sms.12585. Epub 2015 Nov 21. PMID 26589483
- [Background] Jansen JA, Mens JM, Backx FJ, Kolfschoten N, Stam HJ. Treatment of longstanding groin pain in athletes: a systematic review. Scand J Med Sci Sports. 2008 Jun;18(3):263-74. doi: 10.1111/j.1600-0838.2008.00790.x. Epub 2008 Apr 6. PMID 18397195
- [Background] Mosler AB, Crossley KM, Thorborg K, Whiteley RJ, Weir A, Serner A, Holmich P. Hip strength and range of motion: Normal values from a professional football league. J Sci Med Sport. 2017 Apr;20(4):339-343. doi: 10.1016/j.jsams.2016.05.010. Epub 2016 Aug 23. PMID 28185809
- [Background] Serner A, Jakobsen MD, Andersen LL, Holmich P, Sundstrup E, Thorborg K. EMG evaluation of hip adduction exercises for soccer players: implications for exercise selection in prevention and treatment of groin injuries. Br J Sports Med. 2014 Jul;48(14):1108-14. doi: 10.1136/bjsports-2012-091746. Epub 2013 Mar 19. PMID 23511698
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Thorborg K, Tijssen M, Habets B, Bartels EM, Roos EM, Kemp J, Crossley KM, Holmich P. Patient-Reported Outcome (PRO) questionnaires for young to middle-aged adults with hip and groin disability: a systematic review of the clinimetric evidence. Br J Sports Med. 2015 Jun;49(12):812. doi: 10.1136/bjsports-2014-094224. Epub 2015 Jan 13. PMID 25586913
- [Background] Nussbaumer S, Leunig M, Glatthorn JF, Stauffacher S, Gerber H, Maffiuletti NA. Validity and test-retest reliability of manual goniometers for measuring passive hip range of motion in femoroacetabular impingement patients. BMC Musculoskelet Disord. 2010 Aug 31;11:194. doi: 10.1186/1471-2474-11-194. PMID 20807405
- [Background] Holmich P, Uhrskou P, Ulnits L, Kanstrup IL, Nielsen MB, Bjerg AM, Krogsgaard K. Effectiveness of active physical training as treatment for long-standing adductor-related groin pain in athletes: randomised trial. Lancet. 1999 Feb 6;353(9151):439-43. doi: 10.1016/S0140-6736(98)03340-6. PMID 9989713
- [Derived] Alsirhani AA, Muaidi QI, Nuhmani S, Thorborg K, Husain MA, Al Attar WSA. The effectiveness of the Copenhagen adduction exercise on improving eccentric hip adduction strength among soccer players with groin injury: a randomized controlled trial. Phys Sportsmed. 2024 Oct;52(5):497-506. doi: 10.1080/00913847.2024.2321958. Epub 2024 Mar 1. PMID 38376593